CLINICAL TRIAL: NCT05058729
Title: Multiple Sclerosis Partners Advancing Technology and Health Solutions (MS PATHS) - COVID-19 Questionnaire Linkage Sub-Study
Brief Title: MS PATHS COVID-19 Questionnaire Data Linkage Sub-Study
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: US-MSG-11834
Record Dates: First submitted 2021-09-27; First posted 2021-09-28 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Multiple Sclerosis (MS)
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: Participants with multiple sclerosis (MS) or clinically isolated syndrome (CIS) who are enrolled in MS PATHS under Study 888MS001 and have completed at least one COVID-19 questionnaire administered by a participating healthcare institution.

SUMMARY:
The primary objective of this sub-study is to supplement the Multiple Sclerosis Partners Advancing Technology and Health Solutions (MS PATHS) dataset with coronavirus disease 2019 (COVID-19)-related health information obtained from periodic participant questionnaires administered by participating MS PATHS institutions.

ELIGIBILITY:
Key Inclusion Criteria:

1. Be enrolled in MS PATHS under Study 888MS001.
2. Completed one or more COVID-19 questionnaire at a participating MS PATHS institution.
3. Permission for data linkage either obtained when completing a local COVID-19 questionnaire or granted by waiver of informed consent from the local institutional review board (IRB) or ethics committee (EC).

Key Exclusion Criteria:

1. Other unspecified reasons that, in the opinion of the Investigator or Biogen, make the participant unsuitable for participation in the sub-study. A participant only needs to complete the assessments deemed necessary by the Investigator.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with MS or CIS who are enrolled in MS PATHS under Study 888MS001 and have completed at least one COVID-19 questionnaire administered by a participating healthcare institution will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 1507 (Actual)
Dates: Start 2020-12-07 (Actual); Primary Completion 2021-10-08 (Actual); Study Completion 2021-10-08 (Actual)

PRIMARY OUTCOMES:
Number of Completed COVID-19 Questionnaires Able to be Linked to a MS PATHS Participant Identifier (ID) | Up to 17 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (6):
- United States (6):
  - Research Site, Baltimore, Maryland
  - Research Site, St Louis, Missouri
  - Research Site, Las Vegas, Nevada
  - Research Site, New York, New York
  - Research Site, Cleveland, Ohio
  - Research Site, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/